CLINICAL TRIAL: NCT01995461
Title: Effectiveness of Bilateral Transforaminal Epidural Steroid Injections in Degenerative Lumbar Spinal Stenosis Patients With Neurogenic Claudication: A Prospective Outcome Study
Brief Title: Bilateral Transforaminal Epidural Steroid Injections for Degenerative Lumbar Spinal Stenosis
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: biostatistician determined 20 subjects would be adequate to perform statistics
Sponsor: Marshfield Clinic Research Foundation (Other)
Responsible Party: Principal Investigator, Mustafa Farooque, MD, Medical Staff Physician/Clinician, Marshfield Clinic Research Foundation
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: FAR10112
Record Dates: First submitted 2013-11-18; First posted 2013-11-26 (Estimated); Results first posted 2015-11-24 (Estimated); Last update posted 2015-11-24 (Estimated); Status verified 2015-10

CONDITIONS: Spinal Stenosis, Lumbar Region, With Neurogenic Claudication
MeSH Terms: conditions — Spinal Stenosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- BTESI (Experimental): a prospective, non-randomized, case series investigating bilateral transforaminal epidural steroid injections (BTESI)
  Interventions: Drug: bilateral transforaminal epidural steroid injections

INTERVENTIONS:
Drug: bilateral transforaminal epidural steroid injections — BTESI with local anesthetic and steroid, and the use of x-ray contrast, under fluoroscopy guidance performed by the PI. 10mg of dexamethasone (1cc) mixed with 1cc of 2% preservative-free xylocaine (lidocaine) will be injected on each side of the stenotic segment under fluoroscopic guidance after confirming epidural x-ray contrast (1-2cc) spread right before the steroid mixed with local anesthetic injection. The injection may be repeated, but not before 2 weeks after the first injection.
  Other Names: BTESI

SUMMARY:
The most common forms of injection used for the treatment of degenerative lumbar spinal stenosis (DLSS) patients with neurogenic claudication (NC) are the caudal and inter-laminar epidural injections of anesthetic and steroid. Unilateral transforaminal epidural steroid injections (TESI) are also used to alleviate patients' symptoms of NC from DLSS, particularly in patients whose level of stenosis is L4-5 or higher. However, these unilateral injections do not cross the midline, so in cases of lower extremity pain and symptoms on both sides, a bilateral TESI would probably be more beneficial.

To date, there have not been any well designed prospective studies to determine the effectiveness of bilateral TESI below the level of stenosis in DLSS patients with NC. Therefore, the goal of this prospective, non-randomized case-series outcome study is to evaluate the effectiveness of BTESI in alleviating symptoms of NC, as well as improving function in patients with DLSS. The hypothesis is that BTESI at the level below the most stenotic segment of the central canal of the lumbar spine decreases symptoms of NC and improves function in patients with DLSS.

ELIGIBILITY:
Inclusion Criteria:

* Symptoms of back/buttock/leg pain (NOT radicular pain) in a neurogenic claudicatory fashion, relieved by stooping or sitting down, for at least 3 months with no or poor response to conservative treatment (analgesics, NSAIDs, or physical therapy)
* Patients with bilateral buttock and/or bilateral lower extremity pain in a neurogenic fashion with or without lower back pain
* Radiologic documentation of degree of degenerative lumbar spinal stenosis (DLSS)
* MRI/CT showing at least moderate central canal spinal stenosis (neuro-radiologist definition) with symptoms correlating with stenosis (symptoms of back/buttock/leg pain without unilateral radicular pain in a neurogenic claudicatory fashion, relieved by stooping or sitting down)
* Patients choosing to receive BTESI as their next treatment option, following discussions with their spine doctor
* Patients who can give informed consent, could tolerate the procedure, and who are able to understand and answer the forms and questionnaires properly.

Exclusion Criteria:

* Radiologic spinal stenosis without symptoms of spinal stenosis
* Symptoms of neurogenic claudication without at least moderate degree of radiologic spinal stenosis
* Patients with specific lumbo-sacral radicular symptoms or radiculopathy (radicular pain secondary to a single nerve root compression/inflammation; usually follows a specific dermatome in lower extremities; unilateral radiculopathy either from disc herniation or lateral recess stenosis)
* Patients with vascular claudication (pain in the legs secondary to arterial insufficiency)
* Previous lumbo-sacral surgery
* Any condition that does not allow the patient to stand and/or walk for any length of time (e.g., COPD, severe lung disease, etc.)
* Patients with symptomatic hip joint pathology concurrent with spinal stenosis
* A coexisting musculoskeletal condition that would negate functional improvement from the injection (e.g., severe Parkinson disease, hemiparesis, etc.)
* Malignancy or infection to the spine
* Another pain generating condition that would mask the improvement provided by the injection
* Patients who had lumbar epidural steroid injections within the past six months
* Significant psychologic diagnosis and/or dementia
* Patients receiving workman's compensation benefit
* Patients unable to give consent on their own, or who are not able to understand and answer the forms and questionnaires, or their answers will not be reliable.

Ages: 40 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2013-05; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mustafa Farooque, MD, Principal Investigator — Marshfield Clinic/MCRF; James Burmester, PhD, Principal Investigator — Marshfield Clinic Research Foundation
Locations (1):
- Marshfield Clinic, Marshfield, Wisconsin, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | BTESI
Started | 26
Completed | 21
Not Completed | 5
Not completed — Death | 1
Not completed — Lost to Follow-up | 2
Not completed — Withdrawal by Subject | 2

BASELINE CHARACTERISTICS:
Arm/Group | BTESI
Number analyzed (Participants) | 26
Age, Continuous [Median (Full Range); unit: years] | 74.7 [57.7 to 88.1]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14
  Male | 12
Region of Enrollment [Number; unit: participants]
  United States | 26

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline Pain Score at 6 Months
Description: change from baseline (pre-1st injection) pain score, based on a numeric pain scale of 0-10(most severe pain), at 6 months post-1st injection
Time Frame: baseline (pre-1st injection) to 6 months post-1st injection
Measure: Mean (95% Confidence Interval); unit: points
Arm/Group | BTESI
Number analyzed (Participants) | 21
points | -1.6 [-2.9 to -0.2]
Statistical Analysis 1: Comparison: BTESI; Test type: Superiority or Other; p = 0.0252, t-test, 2 sided; paired t-test

2. Secondary Outcome: Change From Baseline Swiss Spinal Stenosis Score at 6 Months
Description: The Swiss spinal stenosis score is a questionnaire composed of 18 multiple choice questions designed to give information as to how the patient's back and leg pain is affecting their ability to manage everyday life. The Swiss spinal stenosis (SSS) questionnaire consists of 12 baseline questions asked of all participants prior to injection and an additional 6 questions asked at each time point post-treatment. The initial 12 questions assess reliability and condition at baseline while the 6 post-treatment questions assess treatment satisfaction. All questions ask the patient to assess symptoms over the previous month with a total maximum score for the initial 12 questions of 53 and a total maximum score of 24 for the 6 additional questions. The final total score is expressed as a percentage of the maximum possible score. Total score increases with worsening disability.
Time Frame: baseline (pre-1st injection) to 6 months post-1st injection
Measure: Mean (95% Confidence Interval); unit: points
Arm/Group | BTESI
Number analyzed (Participants) | 21
points | -8.3 [-14.9 to -1.76]
Statistical Analysis 1: Comparison: BTESI; Test type: Superiority or Other; p = 0.0154, t-test, 2 sided; paired t-test

3. Secondary Outcome: Change From Baseline Oswestry Disability Index at 6 Months
Description: The 2 questions from this Index pertaining to Standing and Walking are being utilized to assess changes in duration of standing and walking in these patients. The two sections of the Oswestry Disability Index (ODI) used in the present study were those related to walking and standing (sections 4 and 6). For each section, the total possible score is 5 and overall ODI score was expressed as a percentage of the maximum possible score (10). Total score increases with worsening disability.
Time Frame: baseline (pre-1st injection) to 6 months post-1st injection
Measure: Mean (95% Confidence Interval); unit: points
Arm/Group | BTESI
Number analyzed (Participants) | 21
points | -7.1 [-14.7 to -1.1]
Statistical Analysis 1: Comparison: BTESI; Test type: Superiority or Other; p = 0.1349, t-test, 2 sided; paired t-test

4. Other Pre Specified Outcome: Change From Baseline Pain Medication Need/Use at 6 Months
Time Frame: baseline (pre-1st injection) to 6 months post-1st injection
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: up to 6 months after injection
Arm/Group | BTESI
Serious Adverse Events (participants affected / at risk) | 0/26
Other Adverse Events (participants affected / at risk) | 0/26

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes